CLINICAL TRIAL: NCT02088801
Title: Phase 2 Study of Evaluation of Videolaryngoscopes in Difficult Airway (SWIVITII)
Brief Title: Evaluation of Videolaryngoscopes in Difficult Airway (SWIVITII)
Acronym: SWIVITII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Lorenz Theiler, Principle investigator, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 106/12_2; SWIVIT II
Record Dates: First submitted 2014-03-11; First posted 2014-03-17 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Difficult Intubation
Keywords: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Airtraq, blade without channel for tracheal tube (Experimental): intubation
  Interventions: Device: Airtraq, blade without channel for tracheal tube intubation
- KingVision , blade without channel for tracheal tube (Experimental): intubation
  Interventions: Device: KingVision , blade without channel for tracheal tube intubation
- A.P. Advance, blade without channel for tracheal tube (Experimental): intubation
  Interventions: Device: A.P. Advance, blade without channel for tracheal tube intubation
- Macintosh (Experimental): intubation
  Interventions: Device: Macintosh

INTERVENTIONS:
Device: Airtraq, blade without channel for tracheal tube intubation — Intubation
  Other Names: Airtraq; A.P. Advance; KingVision; Macintosh
  Arms: Airtraq, blade without channel for tracheal tube
Device: KingVision , blade without channel for tracheal tube intubation
  Arms: KingVision , blade without channel for tracheal tube
Device: A.P. Advance, blade without channel for tracheal tube intubation
  Arms: A.P. Advance, blade without channel for tracheal tube
Device: Macintosh
  Arms: Macintosh

SUMMARY:
In this second phase of the multicenter study the investigators are going to evaluate the use of three different videolaryngoscopes in patients undergoing elective surgery requiring general anesthesia with intubation. The investigators are hypothesizing that these three videolaryngoscopes will succeed for intubation at first attempt in at least 90% of all cases using a difficult airway simulation with extrication collars. As the gold standard, a standard Macintosh blade is being used for comparison.

The study consists of 4 arms. Each arm includes 120 patients, sums up to a total of 480 patients.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery with general anesthesia requiring intubation
* >18 years old
* ASA I-III

Exclusion Criteria:

* known or presumed difficult airway
* risk of pulmonary aspiration
* refusing to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
first attempt intubation success rate | intraoperative

SECONDARY OUTCOMES:
side effects | 1h and 1day after intubation
  sore throat, bleeding, dental injuries

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD MME FERC, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Bern University Hospital and University of Bern, Bern, Canton of Bern, Switzerland